CLINICAL TRIAL: NCT01032525
Title: Epidemiologic Study of Inflammatory Bowel Disease in Monroe County, New York
Brief Title: Monroe County Inflammatory Bowel Disease (IBD) Registry
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: Principal Investigator, Lawrence Saubermann, Associate Professor, University of Rochester
Other Study IDs: 15094
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's Disease; Ulcerative Colitis; IBD; Inflammatory Bowel Disease in Monroe County, NY
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This phase is to register all subjects in Monroe County, New York with Inflammatory Bowel Disease (IBD) not already included to update the database for years 1990-2003. This will give us a truly population based study which will add to our knowledge of IBD epidemiology, allowing us to compare our rates with the rest of the world. We will be able to provide accurate incidence data from 1980 to 2000, and point prevalence from 12/31/2000. It will have special significance because of the relatively stable Monroe County population prior to 2000 (population in 1970=711,917; population in 2000 = 735,343).

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBD who sign consent from 1995-2001

Exclusion Criteria:

* Patients without IBD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of monroe County who had been diagnosed with Crohn's Disease or Ulcerative Colitis
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 1981-01; Primary Completion 2013-05 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
not complete | not complete
  paper is still in progress